CLINICAL TRIAL: NCT01554111
Title: A Randomized Controlled Study Comparing PicoSalax, Versus PicoSalax and Fleet Enema Versus Fleet Enema Alone for Sigmoidoscopy
Brief Title: Comparing Bowel Preparation Regimens for Flexible Sigmoidoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Associate Professor, Queen's University, Department of Medicine, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMED-1429-11
Record Dates: First submitted 2012-03-01; First posted 2012-03-14 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Cathartic Colon
Keywords: Bowel Evacuants; Purgatives
MeSH Terms: interventions — picosulfate sodium; Pico-Salax

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Picosalax with rectal enema (Active Comparator): This arm will receive one satchet of Picosalx and a rectal enema before the sigmoidoscopy for their bowel preparation regimen.
  Interventions: Drug: Pico-Salax and Sodium phosphate enema
- rectal enema (Active Comparator): This group of patients will receive only a rectal enema for bowel preparation before their flexible sigmoidoscopy.
  Interventions: Drug: phosphosoda rectal enema
- Pico-Salax (Active Comparator): patient will take one sachet of pico-salax
  Interventions: Drug: Picosulfate sodium,

INTERVENTIONS:
Drug: Picosulfate sodium, — One sachet of picosalax will be given with at least 4 cups of clear fluids.
  Other Names: PicoSalax
  Arms: Pico-Salax
Drug: phosphosoda rectal enema — The patient will have an enema inserted into the rectum and the liquid contents of the enema will be squeezed into the rectum. The patient will need to hold in the enema for several minutes then can release it.
  Arms: rectal enema
Drug: Pico-Salax and Sodium phosphate enema — Pt will take one sachet of Pico-salax the evening prior to procedure and fleet enema 1 hour before leaving home on the morning of the procedure
  Other Names: Sodium picosulfate
  Arms: Picosalax with rectal enema

SUMMARY:
Objective and Hypothesis:

The investigators objective is to help determine the efficacy of oral and rectal bowel preparation regimens for sigmoidoscopy. The investigators hypothesis is that oral preparation will reduce the amount of repeat rectal enemas required and improve the quality of a bowel exam at the sigmoidoscopy.

DETAILED DESCRIPTION:
Background:

Flexible sigmoidoscopy is an accepted screening modality for colorectal cancer, however, it has put significant strain on endoscopy suite resources. It is important that flexible sigmoidoscopies be done completely and efficiently.

Cleansing before sigmoidoscopy is important to optimize the diagnostic yield of the exam and for polyp detection rates and other colonic lesions. Rectal enemas have been the mainstay of sigmoidoscopy preparations for many endoscopy suites. Procedure prolongation due to the requirement for additional enemas or more washing of a poorly cleansed colon can put a strain on endoscopy time to complete the procedures.

Oral preparations have been a mainstay of colonoscopy cleansing as they allow adequate visualization of the entire colon and are superior to rectal enemas in this regard. Large volume preparations dominate oral colon cleansing. Polyethylene glycol is a large volume solution with an osmotically balanced laxative. Large volume preps are poorly tolerated when compared with small volume preparations. Small volume osmotically active agents can have limitations also, but are being used more frequently with newer agents having a better safety profile.

Few large controlled studies have looked at oral preparation being given in sigmoidoscopy. Tolerability of oral prep has had a negative impact on patient compliance with these regimens in colonoscopy. However, rectal enemas also have had a negative impact on sigmoidoscopy experience.

Many sigmoidoscopies are incomplete or poorly done due to poor prep. Literature for oral bowel preparation regimens has been done predominantly for colonoscopies. The few studies comparing oral preparations to enemas are done without validated methods to record bowel preparation adequately and objectively (1, 2). The goal of our study is to compare the quality of the bowel preparation with oral preparations and rectal enemas to determine which is best.

The investigators plan on determining if the concentration of combustible gases with oral preparations during sigmoidoscopy would be reduced enough to allow for safe electrocautery use during sigmoidoscopy. Hydrogen and methane are two major combustible gases found in a normal colon. These gases can cause explosions in the bowel at the time on sigmoidoscopy if electrocautery is used. The explosive range of hydrogen in air is 4-74%, and for methane this range is 5-15% (3). Levels of combustible gases in the colon have been found to be unsafe in a bowel prepped with two phosphosoda enemas.(4) Several bowel cleansing regimens have been found to be safe for electrocautery by decreasing the concentrations of combustible gases in the colon. Our hypothesis is that a partial oral bowel preparation, will reduce the concentration of combustible gases in the colon to low enough levels to make electrocautery safe during flexible sigmoidoscopy.

Objective and Hypothesis:

Our objective is to help determine the efficacy of oral and rectal bowel preparation regimens for sigmoidoscopy. Our hypothesis is that oral preparation will reduce the amount of repeat rectal enemas required and improve the quality of a bowel exam at the sigmoidoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive male and non-pregnant female patients >18 years old who require outpatient sigmoidoscopy will be considered for inclusion.

Exclusion Criteria:

* previous colorectal surgery and patients with reduced renal function or other medical conditions that would increase the risk of receiving oral PicoSalx would be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Quality of colon cleansing | At the time of the flexible sigmoidoscopy, therefore, within 24 hours of flexible sigmoidoscopy
  The primary outcomes for this trial will be the quality of colon cleansing in the area of the colon examined. We will use a modified Ottawa bowel preparation scoring system measured at the time of endoscopy

SECONDARY OUTCOMES:
Patient tolerance questionnaire | At the time of the flexible sigmoidoscopy, therefore, within 24 hours of flexible sigmoidoscopy
  The questionnaire delivered one half hour prior to the sigmoidoscopy will ask the patient about acceptability of the bowel prep, the patient's compliance with the bowel prep, if the patient would have the same bowel preparation regimen again for another sigmoidoscopy. We also will look at side effects including wind, incontinence, sleep disturbance, bottom soreness, abdominal tenderness, and nausea.
Requirement for an additional rectal enema. | At the time of the flexible sigmoidoscopy, therefore, within 24 hours of flexible sigmoidoscopy
  We also will record whether an additional enema was required to complete an adequate examination.
Maximum length of scope inserted | At the time of the flexible sigmoidoscopy, therefore, within 24 hours of flexible sigmoidoscopy
  The maximum scope length reached during the endoscopic procedure will be recorded. We will also record the type of endoscopic equipment used for the sigmoidoscopy, ie. gastroscope, pediatric colonoscope, sigmoidoscope, etc.
Reason for discontinuing further advancement of the scope | At the time of the flexible sigmoidoscopy, therefore, within 24 hours of flexible sigmoidoscopy
  The main reason for no further advancement of the sigmoidoscope will be recorded as: inadequate prep, patient intolerance, adequate examination length reached for procedure indication.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, MD, Principal Investigator — Queen's University; Samson K. Haimanot, MD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario